CLINICAL TRIAL: NCT05963776
Title: Pulmonary Function Tests Study in Cirrhotic Patients With and Without Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Youssef Mohamed Mahmoud, Resident of Tropical medicine and gastroenterology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-05-02MS
Record Dates: First submitted 2023-06-04; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Complications of Liver Cirrhosis and HCC
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: cases are cirrhotic with hepatocellular carcinoma
  Interventions: Device: spirometry
- control: patients with cirrhosis
  Interventions: Device: spirometry

INTERVENTIONS:
Device: spirometry — pulmonary function tests using spirometry

SUMMARY:
Cirrhosis is a terminal image of chronic liver disease. During the progression from the compensation period to the decompensation period, various complications occur, and the life prognosis is significantly reduced. In recent years, medical treatment for liver cirrhosis has made marked progress. Liver cirrhosis may occur as an end result of manifold infectious, toxic, metabolic, or autoimmune conditions such as viral hepatitis, alcoholism, non-alcoholic steatohepatitis, autoimmune hepatitis (AIH), primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), or a variety of storage disorders such as hemochromatosis, Wilson's disease, and alpha-1-antitrypsin deficiency.

Worldwide, hepatocellular carcinoma (HCC) is a universal problem and its epidemiological data showed variation from place to place. HCC represents the sixth most common cancer worldwide. In Egypt, it represents the fourth common cancer. Egypt ranks the third and 15th most populous country in Africa and worldwide, respectively. HCC is a commonly diagnosed cancer in males and females. It can lead to multi-organ failure including the respiratory system.

Pulmonary function tests (PFTS) are important as an investigation and monitoring of patients with respiratory pathology. They provide important information relating to the large and small airways, the pulmonary parenchyma, and the size and integrity of the pulmonary capillary bed. Although they do not provide a definite diagnosis, different patterns of abnormalities are seen in different respiratory diseases which help to establish the diagnosis.

DETAILED DESCRIPTION:
Cirrhosis is a terminal image of chronic liver disease. During the progression from the compensation period to the decompensation period, various complications occur, and the life prognosis is significantly reduced. In recent years, medical treatment for liver cirrhosis has made marked progress. Liver cirrhosis may occur as an end result of manifold infectious, toxic, metabolic, or autoimmune conditions such as viral hepatitis, alcoholism, non-alcoholic steatohepatitis, autoimmune hepatitis (AIH), primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), or a variety of storage disorders such as hemochromatosis, Wilson's disease, and alpha-1-antitrypsin deficiency .Worldwide, hepatocellular carcinoma (HCC) is a universal problem and its epidemiological data showed variation from place to place. HCC represents the sixth most common cancer worldwide. In Egypt, it represents the fourth common cancer. Egypt ranks the third and 15th most populous country in Africa and worldwide, respectively. HCC is a commonly diagnosed cancer in males and females. It can lead to multi-organ failure including the respiratory system.Patients with liver cirrhosis and HCC are vulnerable to many side effects that reduce their lifetime. One of these side effects is hypoxia resulting from Many conditions which can influence the gas exchange in the lungs. Ascites, pleural effusion, hepatomegaly, and basal lung lobes atelectasis are the most commonly identified causes and can disturb oxygen exchange in a restrictive manner. On the other hand, some side effects of cirrhosis such as hepatopulmonary syndrome or portopulmonary hypertension may make the prognosis worse.Pulmonary function tests (PFTS) are important as an investigation and monitoring of patients with respiratory pathology. They provide important information relating to the large and small airways, the pulmonary parenchyma, and the size and integrity of the pulmonary capillary bed. Although they do not provide a definite diagnosis, different patterns of abnormalities are seen in different respiratory diseases which help to establish the diagnosis.There is no simple mechanism to explain the association between liver disease and hypoxemia and there are probably many factors that have a role in its pathogenesis. Although none of them have been proven as the sole reason, nevertheless ascites, hepatopulmonary syndrome, low albumin levels, anemia, respiratory muscle weakness, and extreme hepatomegaly are still considered among the factors implicated in the pathogenesis of hypoxemia in cirrhosis .Pulmonary complications such as hepatopulmonary syndrome and pulmonary hypertension are observed frequently in these patients. The clinical picture characterized by hypoxemia in absence of primary heart and lung diseases in patients with liver failure is called hepatopulmonary syndrome. In hepatopulmonary syndrome, there is an increase in the alveolar-arterial oxygen gradient and a concomitant dilatation of the intrapulmonary vasculature during the inhalation of room air in addition to liver disease. Varying degrees of pulmonary findings including dyspnea, cyanosis, clubbing, and platypnea due to dilatations in the intrapulmonary vasculature (increase in dyspnea upon the shift from lying to standing position) and orthodeoxia (increase in hypoxia upon the shift from lying to standing position), and hypoxemia are seen in patients with HPS in cirrhotic and HCC patients.In general, PFT is employed to measure lung volumes, bronchial obstruction, gas exchange, lung compliance, and ventilatory capacity. Interstitial lung diseases (ILDs) are characterized by reduced lung volumes (restrictive ventilatory impairment), reduced (static) lung compliance, and reduced diffusing capacity. The pattern of lung function impairments does not allow a specific diagnosis to be made, but rather enables one to assess the presence or absence and the severity of lung involvement. Spirometry is a simple test to measure static lung volumes at rest-slow (inspiratory or expiratory) vital capacity (SVC), forced vital capacity (FVC)-and dynamic volumes-forced expiratory volume in 1 s (FEV1), flow-volume loops

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with liver cirrhosis with and without HCC depending on clinical evidence of stigmata of liver disease (e.g. jaundice, ascites, palmar erythema, spider navi, etc), laboratory data and ultra-sonographic features.

Exclusion Criteria:

* Patients with primary pulmonary pathology.
* Coexisting intrinsic heart disease.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with liver cirrhosis with and without HCC depending on clinical evidence of stigmata of liver disease (e.g. jaundice, ascites, palmar erythema, spider navi, etc), laboratory data and ultra-sonographic features.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary complications of liver cirrhosior or HCC | from 1-9-2023 to 1-9-2024
  assess pulmonary functions impairement and complications due to liver cirrhosis or HCC using spirometer device parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Fukui H, Saito H, Ueno Y, Uto H, Obara K, Sakaida I, Shibuya A, Seike M, Nagoshi S, Segawa M, Tsubouchi H, Moriwaki H, Kato A, Hashimoto E, Michitaka K, Murawaki T, Sugano K, Watanabe M, Shimosegawa T. Evidence-based clinical practice guidelines for liver cirrhosis 2015. J Gastroenterol. 2016 Jul;51(7):629-50. doi: 10.1007/s00535-016-1216-y. Epub 2016 May 31. PMID 27246107
- [Background] Lima B, Martinelli A, Franca AV. [Hepatopulmonary syndrome: pathogenesis, diagnosis and treatment]. Arq Gastroenterol. 2004 Oct-Dec;41(4):250-8. doi: 10.1590/s0004-28032004000400010. Epub 2005 Mar 29. Portuguese. PMID 15806270
- [Background] Przybylowski T, Krenke R, Fangrat A, Nasilowski J, Grabczak EM, Styczynski G, Pruszczyk P, Krawczyk M, Chazan R. Gas exchange abnormalities in patients listed for liver transplantation. J Physiol Pharmacol. 2006 Sep;57 Suppl 4:313-23. PMID 17072060